CLINICAL TRIAL: NCT01751815
Title: The Application of Transcutaneous Electric Nerve Stimulation on Acupoints (Acu-TENS) for Pain Relief During Colonoscopy: a Prospective, Randomized, Placebo-controlled Study
Brief Title: Acu-TENS for Pain Relief During Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2011.442-T
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acu-TENS (Experimental)
  Interventions: Procedure: Acu-TENS
- Placebo-TENS (Sham Comparator)
  Interventions: Procedure: Placebo-TENS

INTERVENTIONS:
Procedure: Acu-TENS — Patients randomized to the experimental group will receive Acu-TENS on acupoints relevant to the treatment of abdominal pain and distension, including Zusanli (stomach meridian ST-36), Hegu (large intestine meridian LI-4), Neiguan (pericardium meridian PC-6), Tianshu (stomach meridian ST-25), and Dachangshu (bladder meridian BL-25).
  Arms: Acu-TENS
Procedure: Placebo-TENS — Patients randomized to the control group will receive placebo-TENS at the same acupoints.
  Arms: Placebo-TENS

SUMMARY:
Background:

Colonoscopy is often regarded as a painful and unpleasant procedure. Transcutaneous Electric Nerve Stimulation on Acupoints (Acu-TENS) is a non-invasive modality that has been used successfully to treat pain of various origins, but few good-quality studies have evaluated its role in treating pain and anxiety during colonoscopy.

Objective:

To investigate the efficacy of Acu-TENS in reducing procedure-related pain and the consumption of sedatives/analgesics during colonoscopy.

Design:

Prospective, randomized, placebo-controlled study.

Subjects:

One hundred and twenty eight consecutive patients undergoing first-time elective day-case colonoscopy without previous experience of acupuncture/Acu-TENS will be recruited.

Interventions:

Patients will be randomized to receive either 45 minutes of Acu-TENS or placebo-TENS before colonoscopy. The acupoints relevant to the treatment of abdominal pain and distension, including Zusanli, Hegu, Neiguan, Tianshu, and Dachangshu will be used. For the placebo-TENS group, a non-conductive plastic film will be placed between the acupoint and the electrode so that no current will be transmitted. Acu-TENS and placebo-TENS will be continued throughout colonoscopy. A mixture of Propofol and Alfentanil, delivered by a patient-controlled syringe pump, will be used for sedation/analgesia in both groups.

Outcome measures:

Primary outcome: doses of patient-controlled sedation/analgesia consumed. Secondary outcomes: pain and satisfaction scores according to a visual analog scale, cecal intubation rate/time, and episodes of hypotension/desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged between 18 and 60 years) undergoing first-time elective day-case colonoscopy
* Patients with American Society of Anesthesiologists (ASA) grading I-II
* Informed consent available

Exclusion Criteria:

* Patients with previous experience of acupuncture or Acu-TENS
* Patients with previous history of colorectal surgery
* Patients who are diagnosed with irritable bowel syndrome according to Rome III criteria
* Patients with chronic pain syndrome
* Patients with psychiatric disorder
* Patients with poor cognitive function
* Patients with renal impairment
* Patients with obstructive sleep apnea syndrome
* Patients with cardiac arrhythmias
* Patients with cardiac pacemaker
* Patients who are pregnant
* Patients who are allergic to the Acu-TENS electrodes or Propofol/Alfentanil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dose of patient-controlled sedation/analgesia consumed | During the procedure (up to 1 day)

SECONDARY OUTCOMES:
Pain score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = no pain, 10 = very painful
Patients' satisfaction score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = not satisfied, 10 = very satisfied
Patients' willingness to repeat the procedure | Up to 1 day
Endoscopists' satisfaction score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = not satisfied, 10 = very satisfied
Cecal intubation rate | During the procedure (up to 1 day)
  Complete colonoscopy is defined as identification of ileocecal valve
Cecal intubation time | During the procedure (up to 1 day)
  The time from introduction of the colonoscope to the cecum
Total procedure time | During the procedure (up to 1 day)
Episodes of hypotension | During the procedure (up to 1 day)
  Defined as systolic blood pressure <90 mmHg
Episodes of desaturation | During the procedure (up to 1 day)
  Defined as SaO2 <90%

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong SAR, China